CLINICAL TRIAL: NCT04990505
Title: Microvascular Injury With Secondary Edema, and Distal Peripheral Vascular Thrombosis Contribution to Clinical Deterioration of Non-critically Ill Patients Hospitalized for SARS-CoV-2 Pneumonia Without Evidence of Pulmonary Embolism: a Preliminary Prospective Observational Study
Brief Title: Microvascular Injury and Distal Thrombosis in COVID-19
Acronym: MIND
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Princesse Grace (Other)
Responsible Party: Sponsor
Other Study IDs: MIND
Record Dates: First submitted 2021-08-03; First posted 2021-08-04 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-02

CONDITIONS: SARS-CoV-2 Infection
Keywords: lung thrombosis; pulmonary embolism; lung scintigraphy; alveolar albumin uptake
MeSH Terms: conditions — COVID-19; Pulmonary Embolism | interventions — Respiration; Perfusion Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: lung ventilation/perfusion scintigraphy — Chest CT-scan will be performed with blocked inspiration.
  Lung ventilation/perfusion scintigraphy imaging will be performed within 24hrs after CT pulmonary angiography, 410MBq of Technegas will be inhaled by patients and ventilation tomography performed thereafter. Then, 185MBq 99mTc-macroaggegates will be injected intravenously followed by the perfusion tomography.
  A combined CT acquisition will be performed.
  The day following lung ventilation/perfusion scintigraphy, 740MBq of Tc99m labeled albumin will be intravenously administered.
  Cardiac gated-blood-pool scintigraphy will be then performed in best septal left anterior oblique and left profile according to specific parameters.
  45-60 min after injection, a non-gated tomographic acquisition over the lungs will be done, with the same parameters than for PS SPECT, resulting in a late albumin acquisition.
  Other Names: Chest CT-scan; CT pulmonary angiography; 99mTc-albumin gated-blood-pool scintigraphy

SUMMARY:
Investigators aimed to better understand the pathophysiology of SARS-CoV-2 pneumonia in non-critically ill hospitalized patients secondarily presenting with clinical deterioration and increase in oxygen requirement

DETAILED DESCRIPTION:
Investigators plan to consecutively enrol 25 patients without clinical or biological evidence for superinfection, without left ventricular dysfunction and for whom a pulmonary embolism was discarded by computed tomography pulmonary angiography. Investigators will investigate lung ventilation and perfusion (LVP) by LVP scintigraphy, and, 24 hours later, left and right ventricular function by 99mTc-labelled albumin gated-blood-pool scintigraphy with late (60 mn) tomographic albumin images on the lungs to evaluate lung albumin retention that could indicate microvascular injuries with secondary edema

ELIGIBILITY:
Inclusion Criteria:

* Non-critically ill patients hospitalized in the COVID-19 Unit of the Centre Hospitalier Princesse Grace of Monaco
* Presenting with a sudden clinical deterioration defined by a respiratory rate impairment and/or a rise of oxygen flow to reach a peripheral capillary oxygen saturation (SpO2) of more than 95% during at least 48 hours
* a diagnosis of pulmonary embolism was discarded by CT pulmonary angiography
* no clinical or biological (procalcitonin levels) evidence of lung superinfection
* without clinical evidence for LV dysfunction

Exclusion Criteria:

* Non confirmed COVID-19 pneumonia according to the WHO guidance by a positive result of RT-PCR assay of nasal and pharyngeal swabs,
* Patients without peripheral pulmonary ground-glass opacities or air-space consolidation on their chest CT scan at admission and common laboratory findings including lymphocytopenia, eosinopenia, significantly elevated markers of organ inflammation such as fibrinogen and C-reactive protein.
* Patients could not be included if their medical condition was unstable or precluded a safe transfer to the nuclear medicine department, if they were under mechanical ventilation (either non-invasive or invasive), if they required critical care unit, or in case of a pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the COVID-19 Unit for SARS-CoV-2 pneumonia with oxygen requirement
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-02-22 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Scintigraphic pattern of peripheral lung thrombosis | During hospitalization
  Determination of the number of patients/pulmonary segments with scintigraphic pattern of peripheral lung thrombosis on the basis of a mismatch between normal ventilation and abnormal perfusion
Pulmonary microvascular injury | During hospitalization
  Determination of the number of patients/pulmonary segments with evidence for microvascular injury on the basis of a lung 99mTc albumin retention, calculated as albumin uptake normalized by the macro-aggregates perfusion uptake

SECONDARY OUTCOMES:
Prognosis evolution at 15 days | 15 days after hospitalization
  Determination of prognosis using categorical variables: worsening or stability vs improvement in the 15 following days, delay to the recovery of a 95% or more SpO2 in ambient air below vs above 15 days, hospitalization duration below vs above 15 days
CT abnormalities prognostic value | 15 days after hospitalization
  The prognostic value of the extent of CT abnormalities, a right ventricular ejection fraction below vs above 50%, a significant albumin uptake (AI/PI) above or equal to 1.7, and the presence and/or number of paradoxically hypoventilated and hypoperfused normal segments will be evaluated by Fisher's exact test and Mann Whitney U test

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maincent C, Perrin C, Chironi G, Baque-Juston M, Berthier F, Paulmier B, Hugonnet F, Dittlot C, Farhad RL, Renvoise J, Serrano B, Nataf V, Mocquot F, Keita-Perse O, Claessens YE, Faraggi M. Microvascular injuries, secondary edema, and inconsistencies in lung vascularization between affected and nonaffected pulmonary segments of non-critically ill hospitalized COVID-19 patients presenting with clinical deterioration. Ther Adv Respir Dis. 2022 Jan-Dec;16:17534666221096040. doi: 10.1177/17534666221096040. PMID 35485327